CLINICAL TRIAL: NCT01074476
Title: Investigation of Oral Glucosamine Effects on Synovial Fluid Viscosity and Viscoelasticity in Osteoarthritis Patients
Brief Title: Effects of Glucosamine on Joint Fluid in Osteoarthritis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H10-00146
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; glucosamine; synovial fluid; viscosity; viscoelasticity; WOMAC
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Glucosamine sulphate tablets
  Interventions: Dietary Supplement: Glucosamine sulphate
- 2 (Placebo Comparator): Placebo tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glucosamine sulphate — 750mg glucosamine sulphate (oral tablets), twice per day for 3 months
  Arms: 1
Other: Placebo — Placebo tablets, twice per day for 3 months
  Arms: 2

SUMMARY:
Osteoarthritis (OA) is the most common joint disease associated with aging. Although many patients take glucosamine supplements as a non-traditional treatment for osteoarthritis, the effectiveness of these supplements is questionable. This study will evaluate glucosamine therapy by directly analyzing two functions of joint fluid that are impaired by osteoarthritis - namely, the abilities to lubricate the joint and absorb shocks during activity. Joint fluid samples will be collected from subjects with knee osteoarthritis and analyzed on a device that simulates typical joint movements. After 3 months of glucosamine supplementation, samples will be collected again to detect potential improvements in joint fluid function.

DETAILED DESCRIPTION:
Background:

The effectiveness of glucosamine sulphate as a treatment for OA is still under debate. Most clinical trials evaluate the effectiveness of OA treatments by self-administered questionnaires about joint pain, stiffness and function (Lequesne Algofunctional Index, Western Ontario and McMaster Universities Osteoarthritis Index - WOMAC).

Although OA has been shown to reduce the viscosity and viscoelasticity of synovial fluid, few studies have used these properties as objective outcome measures in the assessment of glucosamine therapy.

The purpose of this study is to investigate whether glucosamine sulphate oral supplements improve the viscous and viscoelastic properties of synovial fluid in osteoarthritis patients and to explore potential correlations between these properties and subjective assessments of joint pain and function.

Research Method:

Patients will be invited to participate in the study if they have been recommended for synovial fluid aspiration to relieve joint discomfort caused by effusion. Subjects will be randomly assigned to receive either 1500mg of glucosamine sulphate or a placebo daily for 3 months. To relieve pain, subjects will be allowed to take up to 4000 mg of acetaminophen per day. If this is insufficient, NSAIDS will be permitted up to a maximum period of 5 consecutive days. Subjects will be asked to keep a log of their analgesics consumption.

At the baseline visit, patient demographics will be recorded and subjects will be asked to complete the WOMAC index questionnaire, which includes 24 questions to evaluate joint pain, stiffness and physical function. After noting the degree of joint effusion (minor, moderate, severe), an experienced physician will aspirate synovial fluid from the study knee to relieve joint pressure. A sample will be collected for analysis of viscosity and viscoelasticity.

Followup visits will be scheduled after every 4 weeks over the 3-month study period. Each visit will include the completion of a WOMAC questionnaire, clinical assessment of the degree of joint effusion and aspiration of synovial fluid (as necessary) for characterization. Any adverse events (such as headaches, abdominal pain, allergic episodes) will also be reported to the physician.

Changes in synovial fluid viscosity and viscoelasticity will be determined after 3 months of glucosamine supplementation and compared to the placebo group. Correlations between synovial fluid properties and WOMAC scores will also be described.

ELIGIBILITY:
Inclusion Criteria:

* are between 30 and 85 years of age
* are clinically diagnosed with moderate to severe knee OA
* are recommended for synovial fluid aspiration

Exclusion Criteria:

* are clinically diagnosed with inflammatory arthritis
* had previous joint surgery in the study knee
* had injection in the study knee within the past 12 months
* have taken glucosamine and/or chondroitin supplements within the past 3 months

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Changes in synovial fluid viscosity and viscoelasticity compared to baseline | 3 months

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Kwok, Dr, Principal Investigator — University of British Columbia; Dana Grecov, Dr., Study Director — University of British Columbia; Christie Newton, Dr., Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - OASIS Vancouver Clinic, Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - University of British Columbia Health Clinic, Vancouver, British Columbia

REFERENCES:
- [Background] Fam H, Bryant JT, Kontopoulou M. Rheological properties of synovial fluids. Biorheology. 2007;44(2):59-74. PMID 17538199
- [Background] Anadere I, Chmiel H, Laschner W. Viscoelasticity of "normal" and pathological synovial fluid. Biorheology. 1979;16(3):179-84. doi: 10.3233/bir-1979-16306. No abstract available. PMID 508928
- [Background] Schurz J, Ribitsch V. Rheology of synovial fluid. Biorheology. 1987;24(4):385-99. doi: 10.3233/bir-1987-24404. PMID 3663897
- [Background] Vangsness CT Jr, Spiker W, Erickson J. A review of evidence-based medicine for glucosamine and chondroitin sulfate use in knee osteoarthritis. Arthroscopy. 2009 Jan;25(1):86-94. doi: 10.1016/j.arthro.2008.07.020. Epub 2008 Sep 30. PMID 19111223
- [Background] Black C, Clar C, Henderson R, MacEachern C, McNamee P, Quayyum Z, Royle P, Thomas S. The clinical effectiveness of glucosamine and chondroitin supplements in slowing or arresting progression of osteoarthritis of the knee: a systematic review and economic evaluation. Health Technol Assess. 2009 Nov;13(52):1-148. doi: 10.3310/hta13520. PMID 19903416
- [Background] Clegg DO, Reda DJ, Harris CL, Klein MA, O'Dell JR, Hooper MM, Bradley JD, Bingham CO 3rd, Weisman MH, Jackson CG, Lane NE, Cush JJ, Moreland LW, Schumacher HR Jr, Oddis CV, Wolfe F, Molitor JA, Yocum DE, Schnitzer TJ, Furst DE, Sawitzke AD, Shi H, Brandt KD, Moskowitz RW, Williams HJ. Glucosamine, chondroitin sulfate, and the two in combination for painful knee osteoarthritis. N Engl J Med. 2006 Feb 23;354(8):795-808. doi: 10.1056/NEJMoa052771. PMID 16495392
- [Background] Matsuno H, Nakamura H, Katayama K, Hayashi S, Kano S, Yudoh K, Kiso Y. Effects of an oral administration of glucosamine-chondroitin-quercetin glucoside on the synovial fluid properties in patients with osteoarthritis and rheumatoid arthritis. Biosci Biotechnol Biochem. 2009 Feb;73(2):288-92. doi: 10.1271/bbb.80418. Epub 2009 Feb 7. PMID 19202302